CLINICAL TRIAL: NCT01571232
Title: Ozurdex for Treatment of Recalcitrant Diabetic Macular Edema.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retina Macula Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Ron P. Gallemore, Physician and CEO of Retina Macula Institute, Retina Macula Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT-406
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Macular Edema; Non-proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy
Keywords: Macular Edema; DME; PDR; NPDR; Ozurdex; Dexamethasone; Avastin; Bevacizumab
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone; Calcium Dobesilate; Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozurdex (Active Comparator): Patients in this group receive Ozurdex at initial visit and at month 4
  Interventions: Drug: dexamethasone intravitreal implant
- Avastin (Active Comparator): Patients in this group receive Avastin Q1 month for 5 months.
  Interventions: Drug: intravitreal bevacizumab

INTERVENTIONS:
Drug: dexamethasone intravitreal implant — Ozurdex, 0.7 mg intravitreal dexamethasone implant, given at initial visit and at month 4 (visit 5)
  Other Names: Ozurdex
  Arms: Ozurdex
Drug: intravitreal bevacizumab — Avastin, 1.25 mg intravitreal bevacizumab, given at initial visit and Q1month for a total of 5 treatments.
  Other Names: Avastin
  Arms: Avastin

SUMMARY:
The purpose of this study is to test the efficacy of an 0.7 mg intravitreal dexamethasone implant (Ozurdex®) on macular leakage and visual acuity for patients with recalcitrant diabetic macular edema.

DETAILED DESCRIPTION:
This is an open-label, Phase II comparative study of an intravitreal dexamethasone implant versus intravitreal bevacizumab (Avastin) in 20 patients with recalcitrant diabetic macular edema and prior treatment with ≥ 2 intravitreal anti-VEGF injections.

ELIGIBILITY:
Inclusion Criteria:

* Presence of NPDR or PDR as confirmed by fluorescein angiography
* Prior treatment with >= 2 intravitreal anti-VEGF injections but no treatment in last 4 weeks
* < 0.1 LogOCT decrease in macular edema on high resolution OCT between initial visit and following treatment with >= 2 intravitreal anti-VEGF injections
* Age 18 years or older
* ETDRS Visual acuity between 3 and 78 letters (approximate Snellen equivalent of 20/25 to 20/800)
* Ability to provide written informed consent
* Capable of complying with study protocol.

Exclusion Criteria:

* Intraocular injection of steroid medication within prior 3 months
* Evidence of significant geographic atrophy on fluorescein angiography in the opinion of the treating physician
* Concurrent ocular disease (wet AMD, significant ERM, etc) that would limit visual acuity in the opinion of the treating physician
* Prior vitrectomy surgery
* Use of systemic steroids (eg, oral, intravenous, intramuscular, epidural, rectal, or extensive dermal) within 1 month prior to day 1.
* Known history of IOP elevation in response to steroid treatment in either eye that resulted in any of the following: a) = 10 mm Hg increase in IOP in response to steroid injection, or b) IOP = 25 mm Hg and required 2 or more anti-glaucoma medications to keep IOP below 21 mm Hg.
* Patients who are pregnant.
* Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron P Gallemore, M.D, Ph.D, Principal Investigator — Retina Macula Institute
Locations (1):
- Retina Macula Institute, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ozurdex | Avastin
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozurdex | Avastin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (1.8) | 61.2 (2.9) | 62.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Change in Visual Acuity (Number of ETDRS Letters).
Description: The measure the change in ETDRS letters for each treatment group from baseline to 6 months.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ETDRS letters
Arm/Group | Ozurdex | Avastin
Number analyzed (Participants) | 9 | 10
ETDRS letters
  Baseline | 67.8 (3.8) | 71.9 (2.9)
  Final Visit | 69.6 (4.8) | 72.9 (3.4)

2. Primary Outcome: The Change in Central Foveal Thickness (Microns on High Resolution OCT).
Description: The measure the change in central foveal thickness for each treatment group from baseline to 6 months.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: microns
Arm/Group | Ozurdex | Avastin
Number analyzed (Participants) | 9 | 10
microns
  Baseline | 385.9 (43.0) | 341.5 (11.3)
  Final Visit | 305.4 (9.1) | 324.3 (10.9)

3. Secondary Outcome: The Change in Macular Leakage on Fluorescein Angiography From Baseline
Description: To qualitatively assess the change in macular leakage on fluorescein angiography from baseline to 6 months for each treatment arm.
Time Frame: 6 months
Population: Fluorescein angiography data were not collected.
Arm/Group | Ozurdex | Avastin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Change in Mean Macular Sensitivity on Microperimetry From Baseline
Description: To assess the change in macular sensitivity on microperimetry from baseline to 6 months for each treatment arm.
Time Frame: 6 months
Population: One patient in the Ozurdex group withdrew consent, one patient in the Avastin group was lost to follow-up, and results were unattainable for two patients due to imaging difficulties.
Measure: Mean (Standard Error); unit: dB
Groups:
- Ozurdex: Patients in this group receive Ozurdex at initial visit and at month 4 dexamethasone intravitreal implant:
  Ozurdex, 0.7 mg intravitreal dexamethasone implant, given at initial visit and at month 4 (visit 5)
Arm/Group | Ozurdex | Avastin
Number analyzed (Participants) | 8 | 8
dB
  Baseline | 5.6 (2.0) | 10.7 (2.2)
  Final Visit | 7.4 (1.2) | 10.7 (1.5)

5. Secondary Outcome: The Change in Mean Central Amplitude on Multi-focal ERG From Baseline.
Description: To assess the change in mean central amplitude on multi-focal ERG from baseline to 6 months for each treatment arm.
Time Frame: 6 months
Population: One patient in the Ozurdex group withdrew consent, one patient in the Avastin group was lost to follow-up, and results were unattainable for three other patients due to testing difficulties.
Measure: Mean (Standard Error); unit: nV/deg2
Arm/Group | Ozurdex | Avastin
Number analyzed (Participants) | 8 | 7
nV/deg2
  Baseline | 27.8 (4.3) | 34.4 (11.0)
  Final Visit | 40.9 (3.8) | 30.3 (6.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ozurdex | Avastin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ozurdex (N=10) | Avastin (N=10)
Elevated Intraocular Pressure (Eye disorders) | 1 | 0 — Greater than 10 mmHg increase in intraocular pressure from baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No